CLINICAL TRIAL: NCT07297784
Title: The Association Between Problematic Media Use and Postoperative Pain Severity in Pediatric Patients Undergoing Tonsillectomy: An Observational Study
Brief Title: Impact of Problematic Media Use on Postoperative Pain in Children Undergoing Tonsillectomy
Status: Enrolling by invitation | Type: Observational
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, Ali Genc, Assistant professor, Tokat Gaziosmanpasa University
Other Study IDs: 25-MOBAEK-341
Record Dates: First submitted 2025-12-09; First posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Adenotonsillectomy
Keywords: Screen addiction; Problematic media use; Pediatric tonsillectomy; FLACC scale

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pediatric Patients Undergoing Adenotonsillectomy: All participants scheduled for elective adenotonsillectomy will complete the short-form Problematic Media Use Scale (PMUS) in the preoperative period. All patients will undergo a standardized surgical procedure performed by the same surgical team, and postoperative analgesia will be administered according to institutional protocol, consisting of weight-based paracetamol dosing for the first 24 hours.
  Postoperative pain severity will be assessed using the FLACC scale at 1, 6, 12, and 24 hours after surgery.
  The primary aim of this observational study is to evaluate the correlation between PMUS scores and postoperative pain levels in children following adenotonsillectomy.

SUMMARY:
This observational study aims to investigate whether problematic media use is associated with postoperative pain severity in children aged 4-11 years undergoing tonsillectomy. A total of 94 parents who consent to participate and have children within the target age range will be included. Data will be collected using a structured questionnaire covering sociodemographic characteristics, family and child media habits, parental attitudes toward screen use, and the Problematic Media Use Scale (PMUS). Postoperative pain will be assessed using the FLACC scale at multiple time points within the first 24 hours after surgery.

DETAILED DESCRIPTION:
Parents of children aged 4-11 years who agree to participate will be enrolled (n=94). The data collection form includes sociodemographic characteristics of the child and family, media use habits of both the child and parents, parental attitudes toward screen exposure, and the Problematic Media Use Scale (PMUS). All children will undergo a detailed history, physical examination, and routine hematological and biochemical tests. Children with allergies, recent upper respiratory infections, asthma, chronic obstructive pulmonary disease, or those who have received NSAIDs within the past 24 hours will be excluded.

Tonsillectomy indications include recurrent tonsillitis and/or tonsillar hypertrophy. All patients will undergo bilateral tonsillectomy via classical extracapsular dissection under general anesthesia. Hemostasis will be achieved with bipolar cauterization and packing. Postoperatively, oral intake will be restricted for 4 hours, and all patients will receive identical analgesic management consisting solely of paracetamol (10 mg/kg) administered three times daily.

The Problematic Media Use Scale (PMUS) was developed by Domoff et al. in 2017 for children aged 4-11 years to assess problematic digital media use. The Turkish validation of both the long and short forms was conducted by Furuncu in 2019. Based on DSM-5 Internet Gaming Disorder criteria, the scale includes items scored on a 5-point Likert scale, with higher scores indicating more problematic use. The short form of PMUS will be used in this study.

Participants will be categorized into two groups based on PMUS scores. Pain intensity will be evaluated using the FLACC scale at the 1st, 6th, 12th, and 24th postoperative hours. The FLACC scale consists of five behavioral categories (Face, Legs, Activity, Cry, Consolability), scored 0-2 each, with total scores ranging from 0 to 10. A score of 0 indicates comfort, 1-3 mild discomfort, 4-6 moderate pain, and 7-10 severe pain or distress.

Sample size was calculated based on a Type I error of 0.05, power of 0.80, and an expected correlation coefficient of r = 0.30 (low-level association) between problematic media use and pain score. This yielded a required sample of 85 participants. Accounting for approximately 10% attrition, the study aims to enroll 94 children.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 4-11 years
* Scheduled for bilateral tonsillectomy
* Parent/guardian capable of completing questionnaires
* Parent/guardian willing to provide informed consent

Exclusion Criteria:

* Allergy, recent cold/upper respiratory infection
* NSAID use within 24 hours before surgery
* Any condition impairing pain assessment
* Refusal of consent

Ages: 4 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Sample size was calculated based on a Type I error of 0.05, power of 0.80, and an expected correlation coefficient of r = 0.30 (low-level association) between problematic media use and pain score. This yielded a required sample of 85 participants. Accounting for approximately 10% attrition, the study aims to enroll 94 children.
Sampling Method: Non-Probability Sample
Enrollment: 94 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
FLACC pain scores | 1, 6, 12, and 24 hours postoperatively
  The FLACC (Face, Legs, Activity, Cry, Consolability) scale is a validated behavioral pain assessment tool used in pediatric patients who are unable to self-report pain reliably. It consists of five categories:Face, Legs, Activity, Cry, Consolability.
  Each category is scored from 0 to 2, resulting in a total score ranging from 0 to 10, where higher scores indicate more severe pain. Scores are interpreted as follows:
  0: Relaxed and comfortable 1-3: Mild discomfort 4-6: Moderate pain 7-10: Severe pain or significant distress In this study, FLACC scores will be recorded at 1, 6, 12, and 24 hours postoperatively.

CONTACTS AND LOCATIONS:
Locations (1):
- Tokat Gaziosmanpasa University, Tokat Province, Tokat Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The data supporting the findings of this study are available from the corresponding author upon reasonable request. Interested researchers may contact the corresponding author via email and provide a brief description of their intended use.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available starting 6 months after publication and will remain accessible for 5 years